CLINICAL TRIAL: NCT05463341
Title: Evaluating an Intervention to Prevent Overdoses in Rural and Urban Counties
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Nichole Michaels, Principal Investigator, Nationwide Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCH
Record Dates: First submitted 2022-06-01; First posted 2022-07-19 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Opiate Overdose; Fentanyl Overdose; Harm Reduction
MeSH Terms: conditions — Opiate Overdose; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Each participant in the intervention arm will receive one-on-one education on the purpose, benefits, and limitations of fentanyl test strip (FTS) testing and undergo a brief 20-minute FTS educational intervention (including a 2-3-minute video and hands-on demonstrations on how to use FTS). They will also receive a supply of 10 FTS upon enrollment and continued supply upon request throughout the 2-year follow up period.
  Interventions: Behavioral: Fentanyl Test Strips
- Non-Intervention Arm (No Intervention): Fentanyl test strip (FTS) education and a supply of FTS will be offered to participants in the non-intervention arm of the study during the final quarter of year 5.

INTERVENTIONS:
Behavioral: Fentanyl Test Strips — A brief fentanyl test strip (FTS) education intervention will be given to participants at Project DAWN sites in the intervention arm after enrollment and collecting baseline data. It will be offered one-on-one with participants and will include the purpose, benefits, and limitations of FTS testing, and information on how to use FTS, interpret the results, what to do if the FTS is positive, and how to use FTS for different drug delivery methods. Participants will practice and demonstrate use of the FTS, and the short video on how to interpret the FTS will include an on-camera statement on the importance of testing for fentanyl. The video will be accessible to participants after study enrollment. Participants will be advised of the possibility of both false positive/negative results, and that the drugs may be mixed with other substances not detectable with FTS. Participants will be encouraged to practice other harm reduction strategies.
  Arms: Intervention Arm

SUMMARY:
The purpose of the study is to investigate the feasibility, acceptability, and associated benefits and harms of integrating FTS education and distribution into select Project DAWN sites in rural and urban communities in Ohio.

DETAILED DESCRIPTION:
Purpose: Opioid-related fatalities are a leading cause of death in Ohio and nationally, with an increasing number of overdoses attributable to fentanyl. Rapid fentanyl test strips (FTS) test for the presence of some types of fentanyl in urine samples and are increasingly being used to check illicit drugs for fentanyl before they are used. FTS use is a promising harm reduction strategy and research shows when people who use drugs (PWUD) receive a positive result, they are more likely to perform overdose risk reduction behaviors. However, access to FTS is limited, and there are barriers to the adoption of this intervention in some communities. This study will investigate FTS distribution and education as a harm reduction strategy to prevent overdoses among PWUD. Study findings will contribute valuable information about the feasibility and acceptability of integrating FTS drug checking into Project DAWN sites in rural and urban communities in Ohio and help us achieve our long-term goal of reducing overdose deaths.

Study Design: Project DAWN sites that volunteer to participate in the study will be randomly assigned to either the intervention or non-intervention arm of the study.

Clients in the intervention arm of the study will receive:

* One-on-one education on the purpose, benefits, and limitations of FTS testing
* A brief 20-minute fentanyl test strip educational intervention, including a 2-3-minute video and hands-on demonstrations on how to use FTS
* A supply of FTS upon enrollment and throughout the 2-year follow up period

Clients in the non-intervention arm of the study will receive:

• FTS education and a supply of FTS will be offered to participants in the non-intervention arm in the last year of the study

Consent: Written documentation of informed consent will be obtained from all participants.

Incentives: Participants will be compensated for their time with a gift cards for completing the baseline survey, the survey at 6-months, and each biweekly survey.

Recruitment and Retention: Having a close partnership with Project DAWN sites will help us recruit and retain study participants. In addition to key informant interviews in year one and questionnaires in year five, the research team will survey coordinators quarterly to collect data on Project DAWN site and coordinator experiences, identify concerns, and take corrective actions. The investigators will also maintain regular communication with Project DAWN site coordinators when the study staff are onsite.

The research team will handle all enrollment of study clients, delivery of the FTS intervention, and follow up with study participants. Project DAWN sites will be asked to provide a small space for the research team to enroll participants and provide the FTS intervention (if applicable). The sites will also be asked to refer potentially eligible individuals to the research team at times when they are on-site.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Visitor to a Project DAWN site in Ohio that does not currently distribute FTS and has agreed to participate in the study
* Self-reported use of illicit drugs or prescription drugs purchased on the street within the past 6 months
* Has a phone number or email address to allow for follow-up contact
* Understands English (Based on the 2012-2016 American Community Survey, only 2.4% of Ohioans 5 years and older speak English less than "very well.")

Exclusion Criteria:

- None (must meet inclusion criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Determine the perceived barriers and facilitating factors associated with incorporating FTS education and distribution in existing OEND programs in rural and urban counties. | Quarter 2 of Year 1
  Key informant interviews with all site personnel and peer recovery mentors.
  Quantitative Data/Process Measures:
  * # interested Project DAWN sites
  * # Project DAWN sites enrolled
  * # potential participants who request to enroll
  * # participants successfully enrolled
  * # people who receive FTS education and testing materials at baseline
  * # replacement FTS requested/distributed
  * total # FTS distributed
  * proportion of participants in the intervention arm who complete the biweekly surveys
  * proportion of participants who complete the 6-month follow-up questionnaire
Determine the perceived barriers and facilitating factors associated with incorporating FTS education and distribution in existing OEND programs in rural and urban counties. | Quarter 3 of Year 5
  Follow up with intervention arm site personnel to gauge satisfaction with the program and identify any concerns.
  Quantitative Data/Process Measures:
  * # interested Project DAWN sites
  * # Project DAWN sites enrolled
  * # potential participants who request to enroll
  * # participants successfully enrolled
  * # people who receive FTS education and testing materials at baseline
  * # replacement FTS requested/distributed
  * total # FTS distributed
  * proportion of participants in the intervention arm who complete the biweekly surveys
  * proportion of participants who complete the 6-month follow-up questionnaire
Determine the perceived barriers and facilitating factors associated with incorporating FTS education and distribution in existing OEND programs in rural and urban counties. | Quarter 2 of Year 5
  Interview intervention arm site personnel to identify barriers and facilitating factors related to offering FTS education and distribution at OEND sites.
  Quantitative Data/Process Measures:
  * # interested Project DAWN sites
  * # Project DAWN sites enrolled
  * # potential participants who request to enroll
  * # participants successfully enrolled
  * # people who receive FTS education and testing materials at baseline
  * # replacement FTS requested/distributed
  * total # FTS distributed
  * proportion of participants in the intervention arm who complete the biweekly surveys
  * proportion of participants who complete the 6-month follow-up questionnaire
Determine the perceived barriers and facilitating factors associated with incorporating FTS education and distribution in existing OEND programs in rural and urban counties. | 6-month follow-up
  Interview intervention arm sites about the acceptability of the program.
  Quantitative Data/Process Measures:
  * # interested Project DAWN sites
  * # Project DAWN sites enrolled
  * # potential participants who request to enroll
  * # participants successfully enrolled
  * # people who receive FTS education and testing materials at baseline
  * # replacement FTS requested/distributed
  * total # FTS distributed
  * proportion of participants in the intervention arm who complete the biweekly surveys
  * proportion of participants who complete the 6-month follow-up questionnaire
Test the hypothesis that PWUD who receive FTS education and testing materials as part of an OEND program will have improved knowledge and self-efficacy regarding how to test drugs for fentanyl and strategies for lowering their risk of an opioid overdose. | 6-month follow-up
  All participants (in both the intervention and non-intervention arms) will complete a questionnaire at enrollment (for the intervention group, prior to the intervention) and again at 6 months. Both questionnaires (baseline and 6 months) will include the same questions about the participant's knowledge of and self-efficacy in reducing their risk of an opioid overdose by using FTS (Appendix). Participants will be compensated for their time with gift cards for completing the questionnaires.
Test the hypothesis that individuals who receive FTS education and testing materials as part of an OEND program will have a lower opioid overdose rate than individuals who receive OEND only ("usual practice"). | Quarter 3 of Year 5
  Participants in the intervention arm will be contacted biweekly for 2 years and asked if they had an overdose in the past 2 weeks and, if so, what drug they were using at the time. Intervention arm participants will be asked to notify the study team when they receive a positive FTS result. Participants in the non-intervention arm will be contacted biweekly up to a maximum of 2 years after enrollment to ask if they had an overdose in the past 2 weeks and, if so, what drug they were using at the time. Fatal overdoses among participants in the intervention and non-intervention arms of the study will be identified by reviewing death certificates issued by the Ohio Department of Health quarterly starting in Year 2. Participating Project DAWN sites will be asked to advise the study team if they become aware of any fatal overdoses among clients who are enrolled in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Nichole Michaels, PhD, Principal Investigator — Nationwide Children's Hospital, Center for Injury Research & Policy; Gary Smith, MD, DRPH, Principal Investigator — Nationwide Children's Hospital, Center for Injury Research & Policy
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified information on the number of overdoses reported to research staff by study participants and what drug the participant thought they were using at the time will be shared with the Ohio Department of Health's Violence and Injury Prevention Section. Personal stories of potential overdoses averted by use of FTS will be shared in a de-identified form in future trainings.
Time Frame: * Number of overdoses will be shared with ODH throughout the study
  * Personal stories of potential overdoses will be shared with no end-date
Access Criteria: De-identified information will be shared with collaborators or for educational purposes only.

REFERENCES:
- [Derived] Short Mejia A, Smith GA, Fernandez SA, Freisthler B, Grella C, Michaels NL. Evaluating fentanyl test strips as a harm reduction strategy in rural and urban counties: study protocol for a randomized controlled trial. Trials. 2024 Sep 4;25(1):587. doi: 10.1186/s13063-024-08440-y. PMID 39232778